CLINICAL TRIAL: NCT04031365
Title: Acupuncture for Sleep Disturbances in Post-Deployment Military Service Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jane J. Abanes, CDR, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHOK.2019.0055
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias | interventions — Acupuncture Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture and Cognitive Behavioral Therapy (Experimental): Participants will receive four sessions of a brief acupuncture therapy in addition to a brief cognitive behavioral therapy.
  Interventions: Procedure: Acupuncture; Behavioral: Cognitive Behavioral Therapy
- Cognitive Behavioral Therapy (Active Comparator): Participants in this group will receive a brief cognitive behavioral therapy in addition to four telephone follow-ups.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Procedure: Acupuncture — Use of sterile, disposable needles in acupuncture
  Arms: Acupuncture and Cognitive Behavioral Therapy
Behavioral: Cognitive Behavioral Therapy — psychotherapy

SUMMARY:
This randomized study will evaluate the effect of a brief acupuncture therapy in addition to a brief cognitive behavioral therapy in mitigating sleep disturbances in post-deployment military service members using reliable and valid measures.

DETAILED DESCRIPTION:
Introduction: Sleep disturbance is a hallmark symptom of posttraumatic stress disorder (PTSD) and an important antecedent in PTSD recovery in service members who were deployed to Operation Enduring Freedom and Operation Iraqi Freedom. Sleep disturbances (SDs) are important maintainers of PTSD symptoms in service members. Yet, they remain resistant to treatment for many service members. To mitigate the consequences of allostatic load, researchers have investigated the effects of acupuncture as a promising intervention.

Objectives/Aims: The overall goal of this study is to evaluate the effectiveness and perceived benefits of a manual standardized acupuncture (MSSA) as an adjunct therapy to an abbreviated cognitive behavioral therapy (ACBT) in the treatment of SDs in post-deployment military service members. Specific aims include the following: a) To evaluate the effectiveness of MSSA as an adjunct treatment with ACBT, as compared to ACBT alone, for SDs using the Insomnia Severity Index (ISI) and Pittsburg Sleep Quality Index (PSQI) in post-deployment military service members, b) To describe the perceived benefit of MSSA as an adjunct treatment with ACBT, as compared with ACBT alone, for SDs using journal log entries in post-deployment military service members, and c) To explore the influence of participant expectation on the effectiveness of acupuncture on SDs using the Acupuncture Expectancy Scale (AES) in post-deployment military service members in the experimental group.

Methods and Analysis: This is a two-arm, single-center randomized controlled trial in U.S. Naval Hospital, Okinawa, Japan. A random assignment process will be conducted by the primary investigator using permutated block randomization. Service members who meet the study selection criteria and decide to participate will be randomly assigned to either the experimental or control group: 1) Experimental: MSSA and ACBT, or 2) Control: ACBT only and waitlist for acupuncture. Patient-reported questionnaires including ISI, PSQI, and AES will be administered at baseline and then at the completion of the study. Descriptive statistics, reliable change indices, and mixed effects generalized linear models that correct standard errors for repeated assessments will be used to test for the interactive effect of acupuncture treatment and time in the study on each outcome controlling for respective baseline values.

Military Relevance: Given the role of sleep disturbances in posttraumatic stress disorder in the military, intervening early before service members become at risk for severe injuries, hospitalizations, and chronic disability could help decrease burdensome problems.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years of age who have been deployed to operational environments (combat zones, ship deployments, or other austere environments),
2. Self-report of deployment experience and SD symptoms for at least one month,
3. A score of 15 or above on the Insomnia Severity Index (ISI)(C. Morin et al., 2011),
4. A score of 5 or more on the Pittsburg Sleep Quality Index (PSQI)(Buysse et al., 1988),
5. Stable on psychiatric and other medications including blood pressure agents for at least three months,
6. Agrees to participate in a group psychotherapy,
7. Agrees to conduct individual interview via the telephone,
8. Agrees to abstain from sedative-hypnotics and sleep aids including over-the-counter drugs throughout the study (i.e., five weeks), and
9. Able to sign an informed consent.

Exclusion Criteria:

1. Surgery within one month,
2. Substance use disorder diagnosis within one month,
3. Substance use disorder treatment within one month,
4. Pregnant women (acupuncture can result in an induction of labor and spontaneous abortion in rare occasions (White et al., 2008),
5. Has had acupuncture treatment or dry needling (i.e., physical therapy intervention typically utilized for musculoskeletal pain complaints) in the past month,
6. Has had psychotherapy within one month, and
7. Previous diagnosis of other sleep disorders or medical conditions that could impact sleep (e.g., obstructive sleep apnea).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index | 5 weeks
  The ISI is a seven-item standardized self-report questionnaire that measures the subjective symptoms of SDs (C. Morin et al., 2011). These subjective symptoms include the respondents' concerns and distress as a result of problems with sleep. The ISI measure contains seven items including perceived difficulty with sleep-onset, sleep maintenance, and early morning awakenings; satisfaction with sleep patterns; interference of sleep problems with daily functioning; impairment as a result of a sleep problem; and degree of distress or concern with the sleep problem (Bastien, Vallieres, & Morin, 2001). Each item in the ISI is rated from 0 to 4 whereby the higher number indicates more difficulty. The scores are added to yield a range of total scores from 0 to 28 in which a higher score suggests more severe SDs. This scale has good reliability and validity psychometrics and is widely used in research: Cronbach's alpha (0.91), sensitivity (78.1%), specificity (100.0%)(C. M. Morin, 2017).
Pittsburg Sleep Quality Index | 5 weeks
  The PSQI is a 19-item questionnaire that includes seven areas of sleep quality and patterns in adults over the last month including the following components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, SDs, use of sleeping medications, and daytime dysfunction (Buysse et al., 1988). Each item in the scale is scored from 0 to 3 scale (0 = no difficulty; 3 = severe difficulty). The scores are added to yield a global score ranging from 0 to 21 (0 = no difficulty; 21 = severe difficulties in all areas). This scale has good reliability and validity psychometrics and is widely used in research: Cronbach's alpha (0.77 to 0.83), sensitivity (89.6%), specificity (86.5%)(Buysse et al., 1988).

SECONDARY OUTCOMES:
Acupuncture Expectancy Scale | 5 weeks
  Acupuncture Expectancy Scale (AES): The AES is a 4-item questionnaire that measures the participants' expected responses to acupuncture. Participants' expected improvement from acupuncture is rated in a 5-point Likert-type scale ranging from not at all agree to completely agree (Mao et al., 2010). The total possible scores for AES range from 4 to 20, with higher scores indicating greater expectancy. In an initial validation, the instrument's Cronbach's alpha is .82 (Mao et al., 2007). The AES has been found to be reliable, valid, and has acceptable sensitivity to change during treatment starting at week 4 of treatment with increasing statistically significant changes with more acupuncture treatments (Mao et al., 2010).

OTHER OUTCOMES:
Posttraumatic Stress Disorder Checklist | 5 weeks
  The PCL-5 is a 20-item scale that examines the degree of how an individual has been bothered by symptoms associated with a distressing event (Wortmann et al., 2016). Each item is rated from 0 (not at all bothered) to 4 (extremely bothered). Scores are summed to yield a severity score. Permissions to use the PCL-5 are not required (Keane, 1989; Weathers et al., 2013). The PCL-5 scale has good reliability and validity psychometrics (i.e., Cronbach's alpha = 0.75 to 0.95; r = 0.92 to 0.94) (Wortmann et al., 2016) and is widely used in both clinical and research settings.

CONTACTS AND LOCATIONS:
Locations (1):
- U.S. Naval Hospital Okinawa, Okinawa, Japan

REFERENCES:
- [Derived] Abanes JJ, Ridner SH, Dietrich MS, Hiers C, Rhoten B. Acupuncture for Sleep Disturbances in Post-Deployment Military Service Members: A Randomized Controlled Trial. Clin Nurs Res. 2022 Feb;31(2):239-250. doi: 10.1177/10547738211030602. Epub 2021 Jul 6. PMID 34229475
- [Derived] Abanes J, Ridner SH, Rhoten B. Perceived benefits of brief acupuncture for sleep disturbances in postdeployment military service members. J Clin Sleep Med. 2021 Aug 1;17(8):1533-1543. doi: 10.5664/jcsm.9222. PMID 33687323